CLINICAL TRIAL: NCT00657176
Title: A Phase 1, Open-Label, Non-Randomized Study of OPB-31121 in Patients With Advanced Solid Tumors
Brief Title: An Open-Label Phase-1 Study of OPB-31121 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sol Han / Clinical Research Associate, Clinical Research Team
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252-KOA-0701
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OPB-31121 — * 100mg tablet
  * oral administration, Qd

SUMMARY:
This is an open-label, non-randomized, single-center, dose-escalation study in patients with advanced solid tumors. Six dose levels (100, 200, 400, 600, 800, and 1000 mg/day) are planned for the study. In this study, OPB-31121's potential for toxic effects will be evaluated in patients with advanced solid tumors to evaluate the recommended dose for use in subsequent studies. The pharmacokinetics and antitumor effect of the compound will also be investigated.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed solid tumor refractory to standard therapy or for which there is no standard therapy
2. Age: more than 19 years
3. ECOG performance status: less than 2
4. Life expectancy of longer than 3 months
5. Adequate vital organ function as follows:

   * Bone marrow function

     * neutrophils: more than 1,500 per microliter
     * platelets: more than 75,000 per microliter
     * hemoglobin: more than 10.0g per deciliter
   * Hepatic function

     * AST and ALT: less than 2.5 x institutional upper limit normal
     * serum total bilirubin: less than 2.5 x institutional ULN
   * Renal function

     * Serum creatinine: less than 1.5 x institutional ULN
6. Capable of swallowing OPB-31121 tablets
7. Ability to understand and willingness to sign written informed consent document for participation in the trial and for analysis of genotypes CYP2C9 and NAT2
8. No chemotherapy, radiotherapy, surgery, or immunotherapy within 4 weeks prior to study entry and recovered from any prior toxicity

Exclusion criteria:

1. Symptomatic CNS metastasis
2. Uncontrolled concurrent illness, including active infection, heart failure, angina pectoris, and cardiac arrhythmia
3. Psychiatric illness that would limit compliance with study requirements
4. Pregnant or breast-feeding women and women of childbearing potential who cannot or will not use effective contraceptive measures
5. Administration of another investigational agent within 6 months prior to study entry
6. Use of CYP3A4 and CYP2C9 inducers, inhibitors, or substrates, and CYP2B6, CYP2C8 and CYP2D6 substrates
7. Hyperlipidemia:

   Total cholesterol:more than 300 milligram per deciliter or Triglycerides:

   more than 2.5 x institutional ULN
8. Abnormal thyroid function: Hypothyroidism or hyperthyroidism of grade 2 or higher (graded according to the NCI-CTCAE)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Cycle 1

SECONDARY OUTCOMES:
Safety and dose-limiting toxicity | Duration of Study
Pharmacokinetics | Cycle 1
Antitumor effect | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, PhD, Principal Investigator — Division of Hematology and Medical Oncology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea